CLINICAL TRIAL: NCT06769581
Title: The Effect of Dexamethasone Adjuvant to Varying Doses of Bupivacaine on Motor and Sensory Blockade in Infraclavicular Brachial Plexus Blockade
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Döndü Genc Moralar, Assoc. Prof., Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 159
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Infraclavicular Brachial Plexus Block; Dexamethasone Administration; Bupivacaine
Keywords: infraclavicular brachial plexus block; dexamethasone; bupivacaine; concentration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: 0.5% bupivacaine only (Active Comparator): Group 1: 25 ml of 0.5% bupivacaine for infraclavicular brachial plexus block
  Interventions: Procedure: Infraclavicular Brachial Plexus Blocks
- Group 2: 25 ml of 0.5% Bupivacaine and 4 mg Dexamethasone (Experimental): Group 2: 25 ml of 0.5% Bupivacaine and 4 mg Dexamethasone-containing local anesthetic solution for infraclavicular brachial plexus block
  Interventions: Procedure: Infraclavicular Brachial Plexus Blocks
- Group 3: 25 ml of 0.375% Bupivacaine and 4 mg Dexamethasone (Experimental): "Group 3: 25 ml of 0.375% Bupivacaine and 4 mg Dexamethasone-containing local anesthetic solution for infraclavicular brachial plexus block.
  Interventions: Procedure: Infraclavicular Brachial Plexus Blocks
- Group 4: 25 ml of 0.25% Bupivacaine and 4 mg Dexamethasone-containing local anesthetic solution (Experimental): Group 4: 25 ml of 0.25% Bupivacaine and 4 mg Dexamethasone-containing local anesthetic solution for infraclavicular brachial plexus block.
  Interventions: Procedure: Infraclavicular Brachial Plexus Blocks

INTERVENTIONS:
Procedure: Infraclavicular Brachial Plexus Blocks — Lateral sagittal technique infraclavicular brachial plexus block

SUMMARY:
This single-center, prospective, randomized, double-blinded controlled trial investigates the effects of adding 4 mg dexamethasone to different concentrations of bupivacaine on motor and sensory block duration in infraclavicular brachial plexus block. A total of 120 ASA I-II patients aged 18-65 undergoing elective surgeries of the hand, wrist, forearm, or elbow will be randomly assigned to one of four groups:

Group 1: 25 mL of 0.5% bupivacaine. Group 2: 25 mL of 0.5% bupivacaine with 4 mg dexamethasone. Group 3: 25 mL of 0.375% bupivacaine with 4 mg dexamethasone. Group 4: 25 mL of 0.25% bupivacaine with 4 mg dexamethasone. The infraclavicular block will be performed using a lateral sagittal approach under ultrasound and nerve stimulator guidance. Primary outcomes include the duration of motor and sensory block, assessed with a motor block scale and pin-prick sensory test. Secondary outcomes include block onset times, postoperative pain scores (Visual Analog Scale), total analgesic consumption within 48 hours, time to first postoperative analgesic, and rates of rescue block or conversion to general anesthesia.

This study aims to evaluate whether combining dexamethasone with lower concentrations of bupivacaine can maintain block efficacy while reducing local anesthetic dosage, potentially improving the safety and effectiveness of peripheral nerve block protocols.

DETAILED DESCRIPTION:
This study investigates whether adding dexamethasone, a commonly used steroid, to different strengths of bupivacaine (a local anesthetic) can improve the effectiveness and duration of nerve blocks used for upper limb surgeries. The nerve block in this study is an infraclavicular brachial plexus block, which numbs the arm and hand by targeting specific nerves near the shoulder. This type of anesthesia is often preferred for surgeries of the hand, wrist, forearm, or elbow because it reduces pain and the need for general anesthesia.

What Is Being Studied? The research focuses on four groups of patients receiving different mixtures of bupivacaine, with or without dexamethasone. Each patient will receive the same volume of anesthetic solution (25 mL) through a standardized procedure performed under ultrasound and nerve stimulator guidance.

* Group 1: 0.5% bupivacaine only.
* Group 2: 0.5% bupivacaine with 4 mg dexamethasone.
* Group 3: 0.375% bupivacaine with 4 mg dexamethasone.
* Group 4: 0.25% bupivacaine with 4 mg dexamethasone. Why Is This Important? Local anesthetics like bupivacaine can effectively block pain, but using higher concentrations may carry risks, such as muscle weakness or local anesthetic toxicity. Combining dexamethasone with lower concentrations of bupivacaine might extend the block's duration and effectiveness, potentially reducing the total amount of anesthetic needed. This could improve patient safety and recovery while maintaining excellent pain control.

How Will It Be Done? The study involves 120 adult patients aged 18-65, all undergoing elective upper limb surgeries. Participants will be randomly assigned to one of the four groups, and both the patients and the doctors evaluating their progress will not know which group they are in.

Before surgery, each patient will receive the nerve block. The anesthetic solution will be injected near the shoulder, targeting specific nerves with the help of ultrasound and a nerve stimulator. Researchers will measure:

* How quickly the block starts working (block onset time).
* How long the block lasts (motor and sensory block duration).
* The level of pain experienced after surgery, using a pain scale.
* The total amount of pain medication needed within the first 48 hours. What Happens After Surgery? Patients will be closely monitored for pain and block effectiveness. If a patient experiences significant pain during surgery due to an incomplete block, additional anesthetic may be given to the specific nerve, or general anesthesia may be initiated if necessary. Postoperatively, pain relief will be managed with standard medications, and the timing and total dosage will be recorded.

Study Goals:

The primary goal is to determine whether dexamethasone can enhance the duration and effectiveness of the block across different bupivacaine strengths. Secondary goals include understanding how dexamethasone affects block onset time, postoperative pain, and the need for additional pain medications.

Broader Implications:

The findings could help refine anesthesia techniques, making nerve blocks safer and more effective. If lower concentrations of bupivacaine combined with dexamethasone provide similar or better results than higher concentrations alone, this could reduce the risks associated with local anesthetics and improve patient recovery experiences.

This research has the potential to guide future anesthesia practices, benefiting both patients and clinicians by optimizing drug combinations for nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years with ASA I-II who will undergo surgery on the hand, wrist, forearm, or elbow.

Exclusion Criteria:

* Patient refusal to undergo the procedure
* ASA III or higher status
* Diagnosis of diabetes mellitus
* Pregnancy
* History of multiple trauma
* Patients with communication difficulties during or after the procedure
* Sensory impairment at the site of regional anesthesia application
* Presence of a neuromuscular disease
* Open wound or infection at the site of block application
* Coagulopathy that contraindicates the block
* History of allergy to the drugs to be used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Duration of motor and sensory block | 48 hours
  The primary outcome of this study is to examine the effects of different concentrations of bupivacaine combined with dexamethasone, in the same volume, on the duration of motor block and sensory block during infraclavicular brachial plexus block.

SECONDARY OUTCOMES:
Block Onset Time | 30 minutes
  The secondary outcome of this study is the onset time of infraclavicular brachial plexus block.
Postoperative pain levels | 48 hours
  Evaluating the postoperative pain levels in patients. Pain levels will be assessed using the Visual Analog Scale (VAS).
Total analgesic requirements | 48 hours
  Evaluating the total analgesic requirements during the first 48 hours postoperatively.
Block Failure | 30 minutes
  Comparing the rates of rescue blocks and the incidence of conversion to general anesthesia following the administration of infraclavicular brachial plexus block.

CONTACTS AND LOCATIONS:
Overall Officials: Dondu Genc Moralar, Assoc. Prof., Study Director — Gaziosmanpasa Training and Research Hospital
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gupta PK, Hopkins PM. Effect of concentration of local anaesthetic solution on the ED(5)(0) of bupivacaine for supraclavicular brachial plexus block. Br J Anaesth. 2013 Aug;111(2):293-6. doi: 10.1093/bja/aet033. Epub 2013 Mar 26. PMID 23533252
- [Background] Liu J, Richman KA, Grodofsky SR, Bhatt S, Huffman GR, Kelly JD 4th, Glaser DL, Elkassabany N. Is there a dose response of dexamethasone as adjuvant for supraclavicular brachial plexus nerve block? A prospective randomized double-blinded clinical study. J Clin Anesth. 2015 May;27(3):237-42. doi: 10.1016/j.jclinane.2014.12.004. Epub 2015 Jan 28. PMID 25637938
- [Background] Alarasan AK, Agrawal J, Choudhary B, Melhotra A, Uike S, Mukherji A. Effect of dexamethasone in low volume supraclavicular brachial plexus block: A double-blinded randomized clinical study. J Anaesthesiol Clin Pharmacol. 2016 Apr-Jun;32(2):234-9. doi: 10.4103/0970-9185.182108. PMID 27275056